CLINICAL TRIAL: NCT04320667
Title: Phenotype of Urinary CD4+ T Cells as Biomarkers for Prediction of Outcome in ANCA Glomerulonephritis
Brief Title: Urinary T Cell Biomarker for Prediction in ANCA Glomerulonephritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Institute of Health (Other)
Responsible Party: Principal Investigator, Philipp Enghard, PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: ANCAFLURINOCYTE
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Glomerulonephritis Acute
Keywords: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Pauci-Immune Vasculitis; Churg-Strauss Syndrome; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; urinary biomarker; outcome; prediction,; urinary effector memory T lymphocytes; glomerulonephritis; non-invasive biomarker; flow cytometry; treatment outcome; CD4-Positive T-Lymphocytes/immunology
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Churg-Strauss Syndrome; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, lymphocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active ANCA glomerulonephritis: Patients with ANCA related disease (Microscopic Polyangiitis, Granulomatosis with Polyangiitis or Churg-Strauss Syndrome) and active renal involvement
  Interventions: Diagnostic Test: Flow cytometry analysis of urine samples
- Control: Patients with ANCA related disease (MPA, GPA, CSS) without renal involvement or complete remission
  Interventions: Diagnostic Test: Flow cytometry analysis of urine samples

INTERVENTIONS:
Diagnostic Test: Flow cytometry analysis of urine samples — Urine samples will be conserved and frozen upon arrival. All samples will be stained according to T cell and TEC (tubular epithelial cells) panel with fluorochromes.
  T cell panel: CD3, CD4, CD8, CCR7, CD45RO, CD28, CD279; TEC panel: vimentin, cytokeratine, CD10, CD13, CD227, CD326

SUMMARY:
Urinary T lymphocytes may be predictive for clinical outcome in patients with ANCA associated glomerulonephritis (ANCA GN). The investigators hypothesize that the amount of CD4+ effector/memory T cells in urine at time of diagnosis predicts the outcome of patients with active ANCA GN after 6 months of therapy. In a prospective, six-months follow-up study patients' urine will be analysed by flow cytometry every 60 days (+/- 10d). Treatment will be performed to the discretion of the treating clinician. After 6 months of treatment response will be determined as either complete response or partial response.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Biopsy proven ANCA related glomerulonephritis
* In absence of biopsy clinical diagnosis of ANCA related glomerulonephritis

Exclusion Criteria:

* Biopsy proven non-ANCA related kidney disease
* Active menstrual bleeding
* Urinary tract infection
* Kidney transplantation during observational period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at medical wards of Charité Universitätsmedizin Berlin and University College London, The Royal Free Hospital
Sampling Method: Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Phenotype of CD4+ T cells at time point 0 predictive of clinical outcome in patients with active ANCA-assosciated glomerulonephritis | 6 months
  Urinary CD4+ effector/memory T cell counts at time point 0 (time of diagnosis) predict clinical outcome (complete or partial response) after 6 months of treatment in patients with active ANCA-assosciated glomerulonephritis. The frequency of effector/memory CD4+ T lymphocytes is higher in patients with non- or partial response.
  Complete response at 24 weeks: BVAS = 0 Partial response at 24 weeks: at least one renal element of the BVAS score.

SECONDARY OUTCOMES:
Analysis of patients with persistent renal abnormalities as partial response | 6 months
Phenotype of CD8+ T cells at time point 0 predictive of clinical outcome in patients with active ANCA-assosciated glomerulonephritis | 6 months
  Urinary CD8+ effector/memory T cell counts at time point 0 (time of diagnosis) predict clinical outcome (complete or partial response) after 6 months of treatment in patients with active ANCA-assosciated glomerulonephritis. The frequency of effector/memory CD8+ T lymphocytes is higher in patients with non- or partial response.
Subgroup analysis according to treatment | 6 months
Diagnosis of active glomerulonephritis in Patients with ANCA associated vasculitis | 6 months
  Diagnosis according to initial T cell count
Prediction of complete or partial response according to normalization of the amount of urinary T cells at time point 2 and 4 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Enghard, PD Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Charité - Universitätsmedizin Berlin, Berlin, Deutschland, Germany
- The Royal Free London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Enghard P, Rieder C, Kopetschke K, Klocke JR, Undeutsch R, Biesen R, Dragun D, Gollasch M, Schneider U, Aupperle K, Humrich JY, Hiepe F, Backhaus M, Radbruch AH, Burmester GR, Riemekasten G. Urinary CD4 T cells identify SLE patients with proliferative lupus nephritis and can be used to monitor treatment response. Ann Rheum Dis. 2014 Jan;73(1):277-83. doi: 10.1136/annrheumdis-2012-202784. Epub 2013 Mar 8. PMID 23475982
- [Background] Abdulahad WH, Kallenberg CG, Limburg PC, Stegeman CA. Urinary CD4+ effector memory T cells reflect renal disease activity in antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2009 Sep;60(9):2830-8. doi: 10.1002/art.24747. PMID 19714581
- [Background] Lieberthal JG, Cuthbertson D, Carette S, Hoffman GS, Khalidi NA, Koening CL, Langford CA, Maksimowicz-McKinnon K, Seo P, Specks U, Ytterberg SR, Merkel PA, Monach PA; Vasculitis Clinical Research Consortium. urinary biomarkers in relapsing antineutrophil cytoplasmic antibody-associated vasculitis. J Rheumatol. 2013 May;40(5):674-83. doi: 10.3899/jrheum.120879. Epub 2013 Apr 1. PMID 23547217
- [Background] Tomasson G, Grayson PC, Mahr AD, Lavalley M, Merkel PA. Value of ANCA measurements during remission to predict a relapse of ANCA-associated vasculitis--a meta-analysis. Rheumatology (Oxford). 2012 Jan;51(1):100-9. doi: 10.1093/rheumatology/ker280. Epub 2011 Oct 29. PMID 22039267